CLINICAL TRIAL: NCT00637962
Title: Phase I Clinical Trial in Healthy Female Volunteers of Reactogenicity and Immunogenicity of Nine Vaginal Immunisations With HIV CN54gp140 Glycoprotein
Brief Title: Reactogenicity and Immunogenicity of Vaginal CNgp140
Acronym: SG06RS02
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IMP expired prior to completion of recruitment
Sponsor: St George's, University of London (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); York Hospitals (Other)
Responsible Party: Dr David JM Lewis, Chief Investigator, St George's University of London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2007-000781-20; 07/Q0803/29 (Other: Ethical Committee); 2007-000781-20 (EudraCT Number)
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Acquired Immune Deficiency Syndrome
Keywords: HIV; AIDS; Vaccine; intravaginal; mucosal; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active product (Experimental): CN54gp140 + gel
  Interventions: Biological: HIV glycoprotein CN54gp140 (vaccine)
- Gel alone (Placebo Comparator): Gel alone
  Interventions: Biological: Carbopol 974

INTERVENTIONS:
Biological: HIV glycoprotein CN54gp140 (vaccine) — vaginal immunisation with 100ug CN54gp140 antigen in gel on 9 occasions in one menstrual cycle
  Other Names: Previously designated ZM96gp140
  Arms: Active product
Biological: Carbopol 974 — vaginal immunisation with Carbopol 974 P 0.924%; benzyl alcohol 1.09%; sodium hydroxide 0.176%; and purified water 97.81%. alone on 9 occasions in one menstrual cycle
  Other Names: Carbapol gel
  Arms: Gel alone

SUMMARY:
To determine the local (cervico-vaginal) and systemic (whole body) safety of vaginal immunisation with CN54gp140 glycoprotein administered 9 times over a 3 week period.

DETAILED DESCRIPTION:
This randomised, placebo-controlled, double-blind study will primarily assess the local and systemic safety and tolerability of CN54gp140 vaccine. We will also assess whether CN54gp140 vaccine is effective at inducing systemic and/or local specific immune responses.

Thirty healthy women volunteers will be enrolled in this study, at 2 clinical sites. Twenty will receive active CN54gp140 vaccine, and 10 will receive placebo. The placebo group will help us identify side effects caused by CN54gp140. The study is double-blind to eliminate any possibility of researcher or subject bias.

Before administration, CN54gp140 or placebo will be mixed into an aqueous gel vehicle. The treatments will be administered intravaginally in a regimen of 9 immunisations over 3 weeks. Each immunisation of CN54gp140 vaccine will contain 100 µg of CN54gp140 protein, meaning that a total dose of 900 µg will be given to subjects in the active treatment group.

Subjects will be required to make a total of 15 outpatient visits to their local clinical site, over 4 successive menstrual cycles.

Menstrual cycle 1: Screening visits There will be 2 screening visits, at about 4 and 2 weeks before the first immunisation. During these visits the volunteers will be asked questions about their health history and to give permission for us to contact their General Practitioner. Blood and urine samples will be taken for routine laboratory safety tests, and tests for HIV and hepatitis, sexual health, and pregnancy. Blood will also be collected for immunology tests to establish the pre-immunisation state of the immune system. The volunteers will also have a cervico-vaginal examination, and sampling of cervico-vaginal secretions and cells will be done for immunology tests. A photograph of the cervix will be taken to help identify any changes that might occur during the trial. Also, a full medical history and examination will be done.

The volunteers will be given a diary card to take home. They'll be asked to record in the diary any symptoms they have, and medication they take, during the course of the trial. The diaries be regularly checked by the trial staff, who will also make a symptom enquiry at each visit.

Menstrual cycle 2: Immunisation visits There will be 9 immunisation visits, on successive Mondays, Wednesdays and Fridays. The 1st of these visits will be about 7 days after the start of menses. At the 1st, 4th and 9th immunisation visits, blood and urine will be collected for routine laboratory safety and pregnancy tests, and blood collected for immunology tests. Subjects will also have a cervico-vaginal examination, and their temperature, blood pressure and heart rate measured, before self-administering the vaccine.

At the rest of the immunisation visits, subjects will self-administer the vaccine. No other procedures will be done.

Menstrual cycle 3: Sampling visits There will be 3 sampling visits, at about 9, 14 and 21 days after the start of menses. At each visit, subjects will have a cervico-vaginal examination, during which sampling of secretions and cells will be done for immunology tests. Also, blood will be collected for immunology tests, and subjects will have their temperature, blood pressure and heart rate measured. At the 1st and 3rd sampling visits only, blood and urine will be collected for routine laboratory safety tests also.

Menstrual cycle 4: End-of-study visit This visit will be about 10 days after the start of menses. Blood and urine will be collected for routine laboratory safety and pregnancy tests, tests for HIV, and immunology tests. The volunteers will also have a cervico-vaginal examination, during which sampling of secretions and cells will be done for immunology tests, and a full medical examination. A photograph of the cervix will be taken. This visit concludes the subject's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* They are adult female volunteers, 18 to 45 years of age, who have signed an informed consent form following a detailed written explanation of participation in the protocol.
* They are volunteers who are in good health as determined by medical history, physical examination and clinical judgement.
* They are available for the duration of the study.
* They are women who, if capable of becoming pregnant during the study, have agreed to have a pregnancy test immediately before immunisation, and to use appropriate contraception methods during the whole study period. Appropriate contraception shall include physician-prescribed oral hormonal agents, barrier contraceptives, regular and consistent use of condoms without spermicidal agents, or intrauterine devices only. Progesterone-only contraceptives are not suitable due to the lack of a regular menstrual cycle.
* They have agreed not to undertake any vaginal practices other than receptive intercourse with a male or use of sanitary tampons during menses. Use of condoms without spermicidal agents is encouraged.
* They have not donated blood during 3 months prior to study entry and agree to not donate for 3 months after the end of their participation in the study.

Exclusion Criteria:

* They have hypersensitivity to any component of the vaccine used in this study.
* They are found to be HIV antibody or HIV proviral DNA positive at the time of initial screening.
* They have a known or suspected history of cervico-vaginal disease, malignancy or abnormality discovered at time of screening.
* They present in the samples obtained at the screening visit:
* a clinically significant amount of protein or haemoglobin in the urine sample, determined by urine dipstick.
* a clinically significant abnormality in the haematological or biochemical assays.
* Positive tests for Hepatitis B and/or C infection An abnormal value will be defined by the ranges quoted by The Doctors Laboratory for the Vaccine Institute site and Pathology Department, York Hospital for the York site.
* They have a known or suspected impairment of lung, heart, liver, kidney, diseases, blood disorders or immune dysfunction.
* They are receiving immunosuppressive therapy (including systemic steroids).
* They are receiving any medications via vaginal route.
* They have any acute infections (including fever greater than or equal to 38°C) or any chronic disease.
* They present a current problem with substance abuse or with a history of substance abuse which, in the opinion of the investigator, might interfere with participation in the study.
* They have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* They have received an investigational agent within 3 months prior to study entry.
* They cannot speak fluent English, or are planning to leave the area of the study site prior to the end of the study period, or are likely not to complete the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine the local and systemic safety of vaginal immunisation with CN54gp140 glycoprotein administered 9 times over a 3 week period. | 13 weeks

SECONDARY OUTCOMES:
frequency of subjects mounting a cervico-vaginal IgA and IgG response to gp140 after a cycle of 9 vaginal immunisations | 13 wks
frequency of subjects mounting a serum IgG and IgA response to gp140 after a cycle of 9 vaginal immunisations | 13 wks
frequency of subjects with a T-cell response to gp140 in blood after a cycle of 9 vaginal immunisations | 13 wks
frequency of cellular responses to gp140 in cervical cells after a cycle of 9 vaginal immunisations | 13 wks

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's, University of London, UK; Charles Lacey, MD, Principal Investigator — York Hospitals; David JM Lewis, MD, Study Director — St George's, University of London, UK
Locations (2):
- United Kingdom (2):
  - St George's Vaccine Institute, London, England
  - York Hospital, York, England

REFERENCES:
- [Derived] Lewis DJ, Fraser CA, Mahmoud AN, Wiggins RC, Woodrow M, Cope A, Cai C, Giemza R, Jeffs SA, Manoussaka M, Cole T, Cranage MP, Shattock RJ, Lacey CJ. Phase I randomised clinical trial of an HIV-1(CN54), clade C, trimeric envelope vaccine candidate delivered vaginally. PLoS One. 2011;6(9):e25165. doi: 10.1371/journal.pone.0025165. Epub 2011 Sep 30. PMID 21984924
- See also: St George's Vaccine Institute Homepage — http://www.vaccine.ac.uk